CLINICAL TRIAL: NCT05532202
Title: A Mobile Web-Based Parenting Intervention to Strengthen Social-Emotional Development of Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Baggett, Director, Mark Chaffin Center for Healthy Development, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R40MC26822
Record Dates: First submitted 2022-07-23; First posted 2022-09-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Intensive Care Units Neonatal; Parenting; Infant Health
Keywords: Telehealth; Parenting; Infant; Low Birthweight

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Pilot Trial Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants naive to treatment condition and Assessors naive to treatment condition and assessment time point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICU Mom and Baby Net (Experimental): 12-session mobile internet intervention with remote video based coaching targeting maternal mood, sensitive and responsive parenting interactional practices with their infants to facilitate infant social engagement with their mothers. Each session included (1) a web-based self-directed learning program through video-based teaching with check-in questions and provision of immediate corrective feedback, (2) an action plan outlining daily activity practice (homework) based on session content, (3) parent-recorded video and secure upload of session skill practice during interaction with her infant, and (4) a video-based coach call to co-view the parent-recorded video of interaction with her infant.
  Interventions: Behavioral: NICU Mom and Baby Net
- NICU Developmental Awareness System (Active Comparator): Identical to NICU Mom and Baby Net in terms of number of sessions and session structure to serve as an equivalent attention control. 12-session mobile internet intervention with remote coaching of mother awareness of infant developmental milestones. Each session included (1) web-based self-directed learning program through video-based teaching with check-in questions and provision of immediate corrective feedback, (2) an action plan outlining daily activity practice (homework) based on session content, (3) parent-recorded video and secure upload of session skill practice during interaction with her infant, and (4) a video-based coach call to co-view the parent-recorded video of interaction with her infant.
  Interventions: Other: NICU Developmental Awareness System

INTERVENTIONS:
Behavioral: NICU Mom and Baby Net — See arm descriptions.
  Arms: NICU Mom and Baby Net
Other: NICU Developmental Awareness System — See arm description.
  Arms: NICU Developmental Awareness System

SUMMARY:
Low birth weight (LBW) infants are at significantly elevated risk for a host of detrimental outcomes including cognitive, language, and social delays and disabilities, which persist into adulthood. An important protective factor for mitigating risk is sensitive and responsive parenting. While evidence- based home visiting interventions exist and were developed specifically for LBW infants, such as the Play and Learning Strategies program, parents face major obstacles in accessing these interventions. In general, interventions demonstrated to be effective through federal research are very slow to migrate to community service delivery systems. Exacerbating this problem currently is the fact that while VLBW has been increasing, and disproportionately so for those who are poor an of minority status, home visiting programs have sustained some of the largest cuts in their histories. Consequently, there is high demand for effective interventions that can be delivered remotely. Through prior, the investigator team addressed this need by adapting the evidence-based PALS program for web-based delivery using laptop computers with streaming video of in-home parent child interactions and weekly remote coaching. The investigator team then rigorously tested its effects in a sample of low-income mothers and infants with typical birth histories. Results of this randomized controlled study showed pre-post growth in maternal sensitivity behaviors and significant increases in infants' social engagement with their mothers, with moderate to large effect sizes for the intervention group as compared to the control group. These encouraging results provide a strong empirical basis for the enhanced web-based delivery method of the PALS program. Although PALS was originally developed and tested with LBW infants, the web-based version, InfantNet, has not yet been tested with this population. Moreover, emergent trends show that young Latino and Black women most often access the Internet through smart phones, not laptops. Consequently, there is great demand for improving access to evidence-based interventions by making them available on mobile devices such as smart phones. Response: To address the need for more accessible evidence-based interventions, the investigator team will overlay the InfantNet program onto the iPhone and rigorously test its effects with 60 low- income mothers and their LBW infants through a 2-arm, 3 cohort, randomized-controlled design.

DETAILED DESCRIPTION:
Infants born at low birth weight (LBW) present special health care needs and unique challenges to parenting, especially with regard to parents' ability to recognize and sensitively respond to subtle infant social communication signals15. Research has demonstrated the positive impact of parent sensitivity and responsiveness on infant cognitive, social-emotional, and language development as well as subsequent risk mitigation. In contrast, research has demonstrated the negative impact of adverse infant-parent interactions on infant social-emotional difficulties and subsequent internalizing and externalizing disorders. Sadly, poverty and associated environmental risks increase the probability of mothers experiencing both the birth of a LBW infant as well as subsequent parenting difficulties. While targeted interventions can strengthen maternal responsiveness and sensitivity, and, thereby, improve infant social-emotional behavior and developmental outcomes such interventions by and large have yet to reach children and families through home visitation service delivery systems. Moreover, national studies on access to Part-C early intervention programs show that families who are poor and of minority status tend to receive these services later, if at all, and when they do they are more likely to live in communities where service delivery systems are highly stressed and least resourced to deliver effective targeted intervention. Further compounding these service delivery issues is the growing incidence of LBW in the face of historically unprecedented funding cuts to home visitation programs. These issues underscore the need for research examining efficient delivery mechanisms for evidence-based interventions to promote healthy development and early positive behavior for all children, but especially for those with or at risk for disability due to LBW and poverty.

Consistent with the goals of Healthy People 2020 to: (a) achieve health equity, eliminate disparities, and improve the health of all groups; (b) create social and physical environments that promote good health; and (c) promote healthy development and healthy behaviors across every stage of life, we will address Maternal Child Health (MCH) Strategic Research Issue #IV: Promoting the healthy development of Maternal Child Health populations, and its correlate the Maternal Child Health Bureau Strategic Plan Fiscal Years 2003-2007, Goal 2: Promoting an Environment that Supports Maternal and Child Health. We will do so by focusing on efficient delivery of effective prevention strategies aimed at improving health and developmental outcomes for LBW infants. This project builds upon the investigator team's prior National Institute of Mental Health funded research efforts with mothers living in poverty wherein we adapted into a web-based format (InfantNet) the evidence-based Playing and Learning Strategies program (PALS). InfantNet demonstrated success not only in engaging mothers living in disadvantage into the intervention but also significantly strengthening maternal functioning as well as infant behavior in interaction at home13. It is within the context of this prior work and the framework of Healthy People 2020 goals and MCHB investments that the investigator team proposes the following aims and hypotheses: Aim 1: Implement and evaluate the effectiveness of InfantNet for mothers of LBW infants living in societal disadvantage. This aim includes the following: a) Increase the resonance and motivational impact of InfantNet specifically for mothers with LBW infants by adding initial session content related to the special needs of both LBW infants and mothers once exiting the Neonatal Intensive Care Unit (NICU) to go home; and increase the accessibility to LBW-InfantNet for these mothers and infants by overlaying the existing web-based InfantNet program onto mobile web-based access through Smart-Phone delivery, an increasingly prevalent technology in the lives of mothers. The new format will be called NICU Mom and Baby Net; b) Implement a randomized trial to evaluate the impact of NICU Mom and Baby Net with 60 mother-infant dyads living in disadvantage and exiting NICU in the Kansas City inner urban area. Mothers will be randomly assigned to receive either the NICU Mom and Baby Net intervention or a Smart-Phone Attention Control intervention containing information on general infant development. Mothers in both conditions will be provided with an iPhone for mobile web access to their assigned program. Mothers in each condition will be allowed a 6-month intervention period; c) Assess the effectiveness of NICU Mom and Baby Net relative to maternal and infant outcomes. Maternal outcome domains of interest are: observed maternal behavior in interaction with her infant as well as maternal parenting knowledge, attitudes and stress; infant outcome domains of interest are: observed infant behavior in interaction with their mother as well as general infant social-emotional functioning. Outcomes will be assessed at pre- and post-intervention (6-month interval); maintenance on selected outcomes will be assessed again at a 2-month, post intervention follow-up (see Method Variable Table for specific Aim indicators); d) Examine the extent to which maternal satisfaction with and use of the NICU Mom and Baby Net program are associated with positive parent-infant intervention outcomes. Usage indicators will be measured in a formative manner through electronic tracking of usage factors; satisfaction will be measured through within session streaming data report as well as through post-intervention questionnaires (see Variable Table below for specific Aim indicators). Aim 2: Evaluate the extent to which contextual and maternal intrapersonal risks relate to a) initial levels of observed parent and infant behavioral difficulties; and b) parent and infant behavioral change resulting from intervention (see Variables Table). Aim 3: Estimate the preliminary costs associated with InfantNet-VLBW implementation such that the benefits to mothers and their LBW infants can be viewed in relation to these costs by community agencies and policy makers. Hypotheses: 1) Mothers receiving NICU Mom and Baby Net will evidence greater gains in (a) observed maternal sensitive and responsive parenting behavior in interaction with their infant; (b) maternal knowledge of these behaviors; (c) general infant development knowledge; and (d) attitudes towards parenting when compared to their Attention Control Counterparts. Moreover, NICU Mom and Baby Net mothers will evidence greater reductions in: (a) parenting stress when compared to Attention Control mothers. 2) Infants of mothers receiving NICU Mom and Baby Net will evidence greater gains in: (a) observed infant social-emotional behaviors in interaction with their mothers; and (b) general social-emotional functioning when compared to Attention Control infants. 3) Higher levels of initial maternal contextual and intrapersonal risk will not only relate to higher initial levels of observed mother and infant behavioral difficulties, but also act to moderate NICU Mom and Baby Net effects such that those with higher risk levels will evidence lower intervention gain trajectories when compared to lower-risk mothers.

ELIGIBILITY:
Inclusion Criteria:

* Biological or adoptive mothers living in the metropolitan area of Kansas City Missouri
* English speaking
* Infants at birth weighed <2500
* Infants at birth were at least 24 weeks' gestational age,
* Infants were no more than 5 months corrected gestational age at NICU exit

Exclusion Criteria:

* Infant diagnosis of hydrocephalus
* Infant diagnosis bronchopulmonary dysplasia
* Infant diagnosis beyond grade 3 intraventricular hemorrhage
* At the time of screening mother stated she was unable to meaningfully participate due to homelessness, inpatient drug or mental health treatment, physical illness requiring intensive treatment

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Indicator of Parent Child Interaction II- Mother behavior | Assessed Pre-intervention and Post- 6-month intervention
  Pre-post change in direct observation of mother facilitators and interrupters of infant engagement during 5-minute semi-structured free play interaction with infant at home
Indicator of Parent Child Interaction II- Infant behavior | Assessed Pre-intervention and Post- 6-month intervention
  Pre-post change in direct observation of infant engagement and distress behavior during 5-minute semi-structured free play interaction with mother at home

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Baggett, PhD, Principal Investigator — Georgia State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baggett KM, Davis B, Landry SH, Feil EG, Whaley A, Schnitz A, Leve C. Understanding the Steps Toward Mobile Early Intervention for Mothers and Their Infants Exiting the Neonatal Intensive Care Unit: Descriptive Examination. J Med Internet Res. 2020 Sep 22;22(9):e18519. doi: 10.2196/18519. PMID 32960178
- [Background] Davis B, Baggett KM, Patterson AL, Feil EG, Landry SH, Leve C. Power and Efficacy of Maternal Voice in Neonatal Intensive Care Units: Implicit Bias and Family-Centered Care. Matern Child Health J. 2022 Apr;26(4):905-912. doi: 10.1007/s10995-021-03199-z. Epub 2021 Jun 23. PMID 34160758